CLINICAL TRIAL: NCT00525382
Title: A Study Evaluating the Efficacy and Safety of 5 mg Levocetirizine Oral Tablets, Once Daily Versus 10 mg Loratadine Oral Tablets, Once Daily for the Treatment of Chronic Idiopathic Urticaria (CIU)
Brief Title: Study to Compare the Efficacy and Safety Between Levocetirizine and Loratadine for Chronic Idiopathic Urticaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A00334
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2009-09

CONDITIONS: Urticaria
Keywords: Levocetirizine dihydrochloride; Xyzal tablets
MeSH Terms: conditions — Urticaria | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: levocetirizine dihydrochloride

SUMMARY:
Study to Compare the Efficacy and Safety Between Levocetirizine and Loratadine for Chronic Idiopathic Urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 60 years old (inclusive
* having chronic idiopathic urticaria
* at least 6-weeks history of CIU, had at least 3 days of wheals presence/week
* moderate to severe CIU defined as pruritus score ≥ 2, number of wheals ≥ 2, and total symptoms CIU score ≥ 2 at randomization

Exclusion Criteria:

* Asthma requiring daily drug therapy other than ß2 inhaled agonists taken prn
* atopic dermatitis or urticaria requiring an antihistamine treatment or the administration of oral or dermal topical corticosteroids
* urticaria caused by physical factors or other known factors
* cholinergic urticaria
* had urticaria due to other systemic disorders
* were on antihistamine drug currently

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2003-08; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
pruritus severity, assessed by the investigator over 2 weeks of treatment | 2 weeks

SECONDARY OUTCOMES:
Symptom score reducing index; subject severity score at 1 and 2 weeks; investigator global evaluation after 2 weeks of treatment; safety | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma